CLINICAL TRIAL: NCT07180069
Title: Dietary Strategies for Hyperphosphatemia: A Randomized Controlled Study on the Effectiveness of Phosphate-Specific Interventions in Reducing Serum Phosphate Levels in Hemodialysis Patients in a Dialysis Center
Brief Title: Phosphate Diet Strategies to Lower Blood Phosphate in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Hassan Ali Hamzah, Principal investigator, Kufa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of kufa
Record Dates: First submitted 2025-07-20; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Hyperphosphataemia; Phosphorus; Diet Therapy; Chronic Kidney Disease 5D
MeSH Terms: conditions — Hyperphosphatemia | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dietary Advice" (No Intervention): Routine general dietary advice for hemodialysis patients, not phosphate-focused.
- Phosphate-Specific Dietary Education (Other): Individualized dietary education focused on reducing phosphate intake (food choices, portion control, additives).
  Interventions: Other: diet education

INTERVENTIONS:
Other: diet education — Individualized dietary education focused on reducing phosphate intake (food choices, portion control, additives).
  Arms: Phosphate-Specific Dietary Education

SUMMARY:
Raised phosphate levels in the blood (hyperphosphatemia) are frequently observed in hemodialysis patients with chronic kidney failure. In addition to increasing the risk of life threatening complications like heart disease, severe bone disorders, and premature mortality, this condition also poses risks to overall health. Managing phosphate levels effectively is one of the central objectives in treating patients on dialysis.

Control of dietary intake, particularly cutting out high phosphate foods, is one of the most effective ways of managing phosphate levels. Dietary restrictions can be challenging for most patients to adhere to, and effective educational tools for assisting them remain unclear.

This clinical study aims to evaluate the impact of diet-derived education aimed solely at reducing phosphate levels in blood. Patients undergoing hemodialysis at a dialysis center will be randomly assigned to one of two groups. In addition to standard dietary advice, one group will receive targeted phosphate-specific dietary education which includes personalized counseling and aids to encourage selection of low-phosphate foods.

The primary objective is to determine whether participants in the phosphate-specific education group achieve a greater reduction in blood phosphate levels over time as compared to those who receive standard care.

DETAILED DESCRIPTION:
this study occurred from October 2024 to January 2025 at the Hemodialysis Unit in the Department of Nephrology at Al-Sader Medical Teaching Hospital. After screening and applying exclusion criteria, a random sample of 200 hemodialysis patients was selected. They were divided equally into two groups (control and intervention), 100 patients in each group. During the trial, five patients were lost: one opted out, two withdrew due to difficulties complying with the prescribed diet, one was removed while awaiting transplantation, and one succumbed to an infection caused by mucormycosis. Thus, 195 volunteers successfully completed the study trial.

A list of all eligible patients who met inclusion criteria was created. Patients were selected by a simple random sampling method. This method involved assigning each eligible patient a unique identification number and then selecting them randomly using a random number generator tool (Excel). A total of 200 patients were chosen to participate. Selected patients were randomly assigned to either the control or intervention group using a fair randomization method to ensure equal distribution. The researcher flipped a fair coin for each patient: if the coin showed the image face, the patient entered the control group; if it showed the writing face, the patient entered the intervention group, which involved receiving dietary counselling according to the study protocol.

Data were collected using two questionnaires: the Medication Adherence Reporting Scale-5 (MARS-5) and a knowledge about phosphate questionnaire . These tools assessed awareness, dietary habits, and phosphate management. They covered demographic data (age, gender, and educational level), dietary behaviors, and chronic conditions history. Baseline phosphorus, PTH, and calcium (Ca) levels were measured. The study evaluated knowledge of phosphate-rich foods, prior education, and ability to identify high phosphate foods. Awareness of phosphate content in dairy products, canned foods, grains, nuts, and processed meats was assessed. Participants also rated their knowledge, their phosphate intake monitoring, and challenges in reducing phosphate intake (lack of knowledge, food availability, and cost). They further reported whether they received dietary guidance and its clarity. Lastly, the study assessed their perceptions of phosphate management, including its importance in preventing complications and confidence in controlling phosphate levels.

Regular follow-ups were conducted during each dialysis session to monitor adherence. Adjustments were made weekly. Serum phosphate and Ca were measured monthly. October 2024 served as baseline, while November, December, and January 2025 were follow-up points. The control group underwent only baseline data collection without intervention. The intervention included counselling and education for a phosphate-specific diet tailored to each patient's food preferences and eating behavior, maintaining a balanced diet with limited phosphorus (800-1000 mg/day), and simple patient-friendly education about phosphate and Ca physiology, risks of hyperphosphatemia, and high phosphate foods.

Brochures handed out to patients included risks of hyperphosphatemia and lists of foods with high and low phosphate content, as well as additives. Another sheet detailed the amount of phosphorus allowed daily or weekly for each type of food, guidance on regulating phosphorus levels, and the importance of adherence to phosphate binders [Appendix 3]. WhatsApp and telephone calls were used to stay connected with patients, address their inquiries, and ensure they received all necessary information. This approach enabled continuous communication, ongoing support, and monitoring of progress and challenges throughout the intervention period.

As part of the program, food preferences and dietary habits were assessed before assigning meal plans. The primary goal was to ensure that daily phosphorus intake remained within 800-1000 mg/day while maintaining balanced nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-60 years
* Stage 5 CKD patients on hemodialysis
* Receiving ≥2 weekly dialysis sessions for ≥2 months
* Written informed consent provided
* Ability (patient/caregiver) to read, write, and speak Arabic

Exclusion Criteria:

* Age <18 or >60
* Receiving <2 dialysis sessions per week or <2 months duration
* Refusal or inability to provide consent
* Severe mental illness or cognitive impairment
* Acute illness, infection, or hospitalization at enrollment
* Malabsorption conditions or prior GI surgery
* Noncompliance with medication or dialysis regimen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in serum phosphate concentration measured by standard blood test (mg/dL) | Baseline and at weeks 4,8 and week 12
  The primary outcome is the change in serum phosphate level from baseline to 12 weeks. Serum phosphate will be measured using venous blood samples and analyzed with an automated chemistry analyzer in the hospital laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of kufa, Najaf, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT07180069/Prot_SAP_000.pdf